CLINICAL TRIAL: NCT07116382
Title: Risk Factors of Ventilator-Associated Pneumonia in Critically Ill Population of Alexandria; Case-Control Study
Brief Title: Risk Factors of Ventilator-Associated Pneumonia in Critically Ill Population of Alexandria
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, islam elsayed, Researcher, Public Health and Community Medicine Department, Suez Canal University
Other Study IDs: VAPRISK
Record Dates: First submitted 2025-08-02; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Critical Care; Ventilator Associated Pneumonia; Risk Factors
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VAP group: All adult (≥ 18 years) mechanically ventilated patients > 48 hours who are diagnosed with ventilator-associated pneumonia are considered as cases. All possible risk factors for VAP are investigated.
- Matched Control group: Mechanically ventilated (≥ 48 hours) patients and matching with cases regarding their age, gender, and duration of MV. All possible risk factors for VAP are investigated.

SUMMARY:
The aim of the study is to compare cases of ventilator-associated pneumonia with matched controls of mechanically ventilated patients to identify any relevant independent risk factors for ventilator-associated pneumonia. All adult (≥ 18 years) mechanically ventilated patients > 48 hours who are diagnosed with ventilator-associated pneumonia are considered as cases. The control group are mechanically ventilated patients and matching with cases regarding their age, gender, and duration of mechanical ventilation.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia is associated with long hospital stays and significant costs. It also prolongs the length of mechanical ventilation. Incidences of ventilator associated pneumonia are highly influenced by the characteristics of the patient population studied and the criteria and techniques applied for diagnosis. The reported incidence is ranged between 10-20% of mechanically ventilated patients. This incidence in developed countries differs significantly from that in developing ones due to many reasons. Several risk factors are identified. The risk factors can be host, device, or personnel related. The most reproducible risk factor is the duration of mechanical ventilation.

The most well recognized modifiable risk factors are mainly intervention related causes. Despite widespread ventilator-associated pneumonia prevention efforts, there was a 35% increase in the ventilator associated events between 2019 and 2020. Since critically ill patients are dynamic patients who are in need to multiple interventions and techniques, revisiting the risk factors of VAP is essential.

Despite widespread prevention efforts, VAP prevention bundles, surveillance systems and updating definitions by CDC, there was a 35% increase in the ventilator associated events between 2019 and 2020 according to CDC healthcare associated infections progress report in 2020. Since critically ill patients are dynamic patients who are in need to multiple interventions and techniques, revisiting the modifiable risk factors of VAP is essential.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥ 18 years) mechanically ventilated patients > 48 hours who are diagnosed with VAP (Case Group).
* The control group is mechanically ventilated (≥ 48 hours) patients and matched with cases regarding their gender, age, and duration of MV.

Exclusion Criteria:

* Patients with pneumonia prior to MV and those developing pneumonia within 48 hours are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with VAP (cases group) and matched controls without VAP.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
In-ICU mortality | Up to ICU discharge for a maximum of 3 months
  All-Cause Mortality Rate

CONTACTS AND LOCATIONS:
Locations (1):
- AMUH, Alexandria, Egypt